CLINICAL TRIAL: NCT00404222
Title: A Randomized, Multicenter, Single-blind Study Comparing the Analgesic Efficacy and Safety of Extended Release Hydrocodone/Acetaminophen (Vicodin® CR) and Immediate Release Hydrocodone/Acetaminophen (NORCO®) to Placebo in Subjects With Acute Pain Following Bunionectomy
Brief Title: A Study Comparing Vicodin® CR and NORCO® to Placebo in Subjects With Acute Pain Following Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Victor Jorden, MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M05-772
Record Dates: First submitted 2006-11-26; First posted 2006-11-28 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Pain
Keywords: Acute Pain following Bunionectomy
MeSH Terms: conditions — Pain | interventions — Hydrocodone; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- hydrocodone / acetaminophen extended release (Experimental)
  Interventions: Drug: Hydrocodone/Acetaminophen Extended-Release
- Hydrocodone/Acetaminophen Immediate Release (Norco ®) (Active Comparator)
  Interventions: Drug: Hydrocodone/Acetaminophen Immediate Release (NORCO®)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocodone/Acetaminophen Extended-Release — 2 tablets x 1
  Other Names: hydrocodone / acetaminophen extended release
  Arms: hydrocodone / acetaminophen extended release
Drug: Hydrocodone/Acetaminophen Immediate Release (NORCO®) — 1 tablet q 4 hours x 3
  Arms: Hydrocodone/Acetaminophen Immediate Release (Norco ®)
Drug: Placebo — q 4 hours x 3
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness (level of pain control) and safety of the administration of Extended Release Hydrocodone/Acetaminophen and Immediate Release Hydrocodone/Acetaminophen with placebo over a 12 hour dosing period in patients who have had a bunionectomy, and to assess the safety of the drug for 7 days after patients are discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18 to 65
* Scheduled to undergo primary, unilateral, first metatarsal osteotomy (bunionectomy)
* Must meet specific pain intensity criteria on the morning after surgery
* Willing to remain at the study center 2 days following surgery
* If female, must be of non-child bearing potential or practicing birth control

Exclusion Criteria:

* Is allergic to or has a serious reaction to hydrocodone, hydromorphone, oxycodone, acetaminophen, ketorolac, lidocaine, bupivacaine, or mepivacaine
* Is allergic to or has a serious reaction to aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs)
* Has a history of or currently has any active seizure disorder
* Has a history of or any disease causing severe gastrointestinal narrowing or slowing down the gastrointestinal tract
* Has been diagnosed with cancer within the past 3 years
* Requires treatment with certain drugs for depression or psychiatric disorders
* Has specific clinically significant illnesses or laboratory abnormalities
* Received corticosteroid treatment or any investigational drug within a specific timeframe.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-11; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the time-interval weighted sum of pain intensity difference (SPID) using the visual analog scale (VAS) for the 0 to 12 hours following study drug administration. | 12 hours
Sum of Pain Intensity Difference using a 100mm Visual Analog Scale (VAS) | 12 hours

SECONDARY OUTCOMES:
Time-interval weighted sum of pain relief (TOTPAR) | 12 hours
Time-interval weighted sum of pain relief and pain intensity difference (SPRID) | 12 hours
Time to first noticeable pain relief (i.e., onset of pain relief) | 12 hours
Time to first meaningful pain relief (i.e. 50% reduction in pain from baseline) | 12 hours
Proportion of subjects experiencing meaningful pain relief after dosing | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rita Jain, MD, Study Director — Abbott